CLINICAL TRIAL: NCT05159180
Title: Desarrollo de un Nuevo Sistema de Mapeo de Impedancia Para la ablación de Las Arritmias Auriculares en Pacientes
Brief Title: Development of a New Impedance Mapping System for Ablation of Atrial Arrhythmias in Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-IMS-2021-74
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation and Flutter; Atrial Arrhythmia; Atrial Fibrillation Recurrent
Keywords: impedance spectroscopy; phase angle; impedance magnitude; Electroanatomical mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with atrial arrhythmias undergoing catheter ablation of these: Patients will be submitted to mapping of both voltage and tissue impedance. The accuracy of the two maps identifying the extent and transmurality of the infarction will be assesssed by gadolinium imaging.
  Interventions: Device: cardioz mapping

INTERVENTIONS:
Device: cardioz mapping — Patients will be submitted to mapping of both voltage and tissue impedance.

SUMMARY:
Precise identification of the atrial fibrosis is essential for successful catheter ablation of atrial arrhythmias in patients with atrial fibrillation. Voltage mapping of endocardial electrograms is currently used to delineate the anatomical substrate, but this is influenced by the direction of the activation wave front and is limited by the patient-specific thresholds. Mapping of local myocardial electrical impedance may overcome these limitations.

DETAILED DESCRIPTION:
Clinical series: Patients with atrial arrythmias undergoing catheter ablation of these will be submitted to mapping of both voltage and tissue impedance. Likewise, the accuracy of the two maps identifying the extent of the substrate will be assesssed by gadolinium imaging. The impedance system is already constructed and certified for clinical research use.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years.
* That they understand and sign the informed consent.
* That they do not present any contraindication.- Pass the exploration and tests prior to bioimpedance measurements.

Exclusion Criteria:

* Age outside the range described in the inclusion criteria.
* Subjects who present any type of complication during the procedure.
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial arrhythmias undergoing catheter ablation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-12-13 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparative detection of atrial scar by voltage mapping | 30 minutes
  Voltage will be measured at different sites of the atrial scar and healthy tissue.
Comparative detection of atrial scar by impedance mapping | 30 minutes
  Myocardial local impedance spectroscopy will be measured at different sites of the atrial scar and healthy tissue.
Comparative detection of atrial scar by gadolinium enhanced MR imaging | 30 minutes
  Intensity of gadolinium will be measured at different sites of the infarct scar and healthy tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Amoros-Figueras G, Jorge E, Garcia-Sanchez T, Bragos R, Rosell-Ferrer J, Cinca J. Recognition of Fibrotic Infarct Density by the Pattern of Local Systolic-Diastolic Myocardial Electrical Impedance. Front Physiol. 2016 Aug 31;7:389. doi: 10.3389/fphys.2016.00389. eCollection 2016. PMID 27630580
- [Result] Amoros-Figueras G, Jorge E, Alonso-Martin C, Traver D, Ballesta M, Bragos R, Rosell-Ferrer J, Cinca J. Endocardial infarct scar recognition by myocardial electrical impedance is not influenced by changes in cardiac activation sequence. Heart Rhythm. 2018 Apr;15(4):589-596. doi: 10.1016/j.hrthm.2017.11.031. Epub 2017 Dec 27. PMID 29197656
- [Result] Jorge E, Amoros-Figueras G, Garcia-Sanchez T, Bragos R, Rosell-Ferrer J, Cinca J. Early detection of acute transmural myocardial ischemia by the phasic systolic-diastolic changes of local tissue electrical impedance. Am J Physiol Heart Circ Physiol. 2016 Feb 1;310(3):H436-43. doi: 10.1152/ajpheart.00754.2015. Epub 2015 Nov 25. PMID 26608340
- [Derived] Amoros-Figueras G, Moreno-Weidmann Z, Mendez-Zurita F, Soriano-Amores M, Bragos R, Rosell-Ferrer J, Guerra JM. Local multifrequency impedance changes after radiofrequency ablation in human atria: potential use for tissue characterization. Front Cardiovasc Med. 2025 Oct 7;12:1668533. doi: 10.3389/fcvm.2025.1668533. eCollection 2025. PMID 41126919